CLINICAL TRIAL: NCT05079646
Title: An In Vitro Evaluation of Fracture Resistance of Endodontically Treated Teeth Restored With New Contemporary Core Build-up Materials: A Randomized Control Trial
Brief Title: An In Vitro Evaluation of Fracture Resistance of Endodontically Treated Teeth Restored With New Contemporary Core Build-up Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Mahreen Daud, Principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MDaud
Record Dates: First submitted 2021-09-22; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Fracture Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group 1, subgroup A (blue color coded) (No Intervention): Normal teeth with no cavity preparation and no endodontic procedure.
- Group 1, subgroup B (pink color coded) (Experimental): Teeth specimens in which endodontic procedure will be performed and coronal restoration will be done with Zirconomer (shofu).
  Interventions: Other: class 1 and class 2 cavity preparation and restored with contemporary materials
- Group 1, subgroup C (green color coded) (Experimental): Teeth specimens in which endodontic procedure will be performed and coronal restoration will be done with Cention-N (Ivoclar vivodent)
  Interventions: Other: class 1 and class 2 cavity preparation and restored with contemporary materials
- Group 1, subgroup D (black color coded) positive control group (Active Comparator): Teeth specimens in which endodontic procedure will be performed and coronal restoration will be done with Aristaloy Amalgam (Cookson)
  Interventions: Other: class 1 and class 2 cavity preparation and restored with contemporary materials
- Group 2, Subgroup A (Blue color coded) negative control group (No Intervention): Normal teeth with no cavity preparation and no endodontic procedure.
- Group 2, Subgroup B (pink color coded) (Experimental): Teeth specimens in which endodontic procedure will be performed and coronal restoration will be done with Zirconomer (shofu) by using tofflemire retainer and matrix band.
  Interventions: Other: class 1 and class 2 cavity preparation and restored with contemporary materials
- Group 2, Subgroup C (green color coded) (Experimental): Teeth specimens in which endodontic procedure will be performed and coronal restoration will be done with Cention-N (Ivoclar vivodent) by using tofflemire retainer and matrix band.
  Interventions: Other: class 1 and class 2 cavity preparation and restored with contemporary materials
- Group 2, Subgroup D (black color coded) (Active Comparator): Teeth specimens in which endodontic procedure will be performed and coronal restoration will be done with Aristaloy Amalgam (Cookson) by using tofflemire retainer and matrix band.
  Interventions: Other: class 1 and class 2 cavity preparation and restored with contemporary materials

INTERVENTIONS:
Other: class 1 and class 2 cavity preparation and restored with contemporary materials — class 1 and class 2 cavities prepared in extracted teeth after endodontic procedure and then these cavities were filled with new contemporary core buildup materials.
  Arms: Group 1, subgroup B (pink color coded); Group 1, subgroup C (green color coded); Group 1, subgroup D (black color coded) positive control group; Group 2, Subgroup B (pink color coded); Group 2, Subgroup C (green color coded); Group 2, Subgroup D (black color coded)

SUMMARY:
Endodontic treatment is performed frequently which often results in weakening of tooth structure. Coronal restoration is done to restore these endodontically treated teeth. Posts have been used to retain the coronal restoration and reinforce these teeth but unfortunately posts placement results in further weakening of tooth structure. Newer contemporary core buildup materials will be used to restore coronal part of tooth without using endodontic posts and then the fracture resistance of these teeth will be evaluated.

This study will be performed to evaluate the fracture resistance of endodontically treated teeth restored with newer contemporary core buildup materials.

80 recently extracted single rooted caries-free and unrestored premolars will be taken and mounted in acrylic resin blocks. Roots of teeth will be covered with light bodies of condensation silicone impression material to simulate periodontal ligaments. Class 1 and class 2 cavities will be prepared and endodontic treatment will be performed in these teeth specimens. Coronal restoration will be done with three core buildup materials (Cention-N, Zirconomer and Aristaloy Amalgam). Teeth specimens are then divided into group 1 and group 2 (class 1 cavity preparation and class 2 cavity preparation respectively) and each group is further divided into four subgroups: Subgroup A: Control group Subgroup B: Cavities restored with Zirconomer (Shofu) Subgroup C: Cavities restored with Cention-N (Ivoclar vivodent) Subgroup D: Cavities restored with Aristaloy Amalgam (Cookson) Fracture resistance of endodontically treated teeth restored with different core buildup materials will be tested by the Universal testing machine.

DETAILED DESCRIPTION:
Total 80 recently extracted single rooted lower second premolars, extracted for orthodontic treatment, will be selected for this study. Because lower second premolars are commonly extracted for orthodontic purposes and during mastication, the anatomic shape ofpremolars create tendency for separation of cusps. Indenter contacts the tooth and acts as a wedge between buccal and lingual cusps and decrease mean fracture resistance values. So the application of force vertically on cusp inclines found to be appropriate to simulate intraoral clinical conditions.

Teeth will be washed under running water and any soft tissue attached to root surfaces will be scraped off with hand scaler. Teeth disinfected with 0.1% thymol solution and will be stored in 10% formalin solution for four days atleast, until they are used, teeth will be stored in 0.9% saline solution at room temperature.

With the help of computer generated software, Teeth will be randomly divided into two groups. Each group contains 40 teeth. Class 1 cavity preparation will be done in teeth of group 1 with straight fissure diamond bur (HiCare ISO. 109/010) in high speed handpiece (Nsk, Japan) along with water coolant and cavity will be prepared on occlusal fissures.

Intercuspal distance and mesio-distal dimension of teeth will be measured with digital caliper. The buccolingual width of class 1 cavity will be one-third of the distance between buccal and lingual cusps and mesiodistal width would be one-third of mesio-distal distance. Buccal and lingual walls will be parallel to one other and cavo-surface angle of approximately 90 degree will be prepared. Class 2 cavity will be prepared in teeth of group 2, in the same way as class 1 except that proximal box will also be prepared in class 2. The width of occlusal isthmus will be the one-third of intercuspal distance and the buccolingual dimension of approximal preparation will be the one-third of buccolingual dimension of overall crown. Gingival extent of this approximal preparation will be 1mm coronal to cemento-enamel junction and the gingival width would be of 2 +/- 0.2mm. Buccal and lingual walls of occlusal preparation will be parallel to each other.

Class 1 and class 2 cavities are prepared because occlusal and proximal surfaces of teeth are the main surfaces which are subjected to higher forces during mastication and these two surfaces are more susceptible to caries attack and standard method for access opening is from occlusal and proximal surface (if carious lesion involve proximal surface too).

Access cavity for endodontics will be prepared with diamond round bur (HiCare ISO.

001/010). The working length will be taken by introducing the #10 K-file (Mani) in the canal until it becomes visible from apical foramen, The working length will be determined by subtracting 1mm from this estimated length. Endodontic procedure will be carried out in all teeth specimens by using rotary Protaper files (Densply). Sequence of S1, S2 and then F1 and F2 will be followed to prepare the canals at the working length. Canals will be irrigated thoroughly after every file with 2.5% NaOCl solution. After cleaning and shaping, canals will be dried with paper points and obturation will be done with sealer (Sealapex, SybronEndo-Kerr, Glendora, CA, USA) and F2 gutta percha cone (Densply).

Modeling wax will be melted and root of tooth will be dipped in it below cement-enamel junction, this will produce a layer of 0.2 to 0.3 mm of wax on root surfaces. This thickness of wax on root surfaces will be representative to the thickness of periodontal ligament. Teeth will be placed in acrylic resin block of 3cmx 2.5cm such that 1.0 mm of root below cement-enamel junction will be out of the block to simulate the biologic width. Wax will be used as spacer between root and acrylic resin block and will be removed. Light body of condensation silicone impression material will be mixed and poured into resin block. Teeth will be reinserted into acrylic resin blocks with the silicone impression material, which will simulate periodontal ligament. Since the PDL acts as an effective support during the masticatory function and absorb and transmit forces between teeth and alveolar bone. So, to produce the clinical situation and to provide a more accurate assessment of fracture resistance of teeth, teeth are embedded in light body of condensation silicone impression material.

Now, Each group will be randomly divided into four sub-groups. In each sub-group, there will be 10 teeth specimens. To make identification of specimens, each group and sub-group will be color coded. There will be one positive control group and one negative control group among the four subgroups and rest 2 sub-groups will be restored with new contemporary core buildup materials.

GROUP 1 (Yellow color coded) Class 1 cavity preparation

Sub-groups

A (Blue color coded) negative control group: Normal teeth with no cavity preparation and no endodontic procedure.

B (Pink color coded): teeth specimens in which endodontic procedure was performed and coronal restoration was done with Zirconomer (Shofu) C (Green color coded) : teeth specimens in which endodontic procedure was performed and coronal restoration was done with Cention-N (Ivovclar vivodent) D (Black color coded) : teeth specimens in which endodontic procedure was performed and coronal restoration was done with Aristaloy Amalgam (cookson)

GROUP 2 (Purple color coded) Class 2 cavity preparation

Sub-groups

A (Blue color coded) negative control group: Normal teeth with no cavity preparation and no endodontic procedure B (Pink color coded): teeth specimens in which endodontic procedure was performed and coronal restoration was done with Zirconomer (Shofu) by using tofflemire retainer and matrix band.

C (Green color coded) : teeth specimens in which endodontic procedure was performed and coronal restoration was done with Cention-N (Ivovclar vivodent) by using tofflemire retainer and matrix band.

D (Black color coded) : teeth specimens in which endodontic procedure was performed and coronal restoration was done with Aristaloy Amalgam (cookson) by using tofflemire retainer and matrix band.

Each tooth specimen will be individually tested in the Universal testing machine (UTM, INSTRON - 4301 Sr. # H1853, PCSIR Karachi). Tooth specimen will be placed in the holding slot that will be attached to the lower part of testing machine. Rounded stainless steel probe of diameter 6mm will be attached to the upper part of machine. Since, We are evaluating the fracture resistance of tooth that whether the new contemporary material enhances the fracture resisting ability of tooth, the probe will contact the inclined planes of facial and lingual cusps of tooth beyond the margins of restoration. The force will start from 'zero' Newton and then indenter will apply the increasing compressive loads to the inclined planes of buccal and lingual cusps until the tooth fractures and final force (Newtons) will be noted. The applied load would be parallel to the long axis of teeth. Load will be applied at crosshead speed of 1mm/min and will be increased gradually until fracture occurs. Maximum force required to fracture the tooth will be recorded in Newtons.

All sample preparation will be done by the principle investigator and sample testing and scoring will be done by a blinded examiner.

ELIGIBILITY:
Inclusion Criteria:

* Teeth extracted from the age group of 18-30 years
* Single rooted lower 2 nd premolars
* Sound teeth with no caries

Exclusion Criteria:

* Incompletely closed apices
* Root resorption, fracture, or craze lines
* Endodontically treated or restored teeth

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
fracture resistance (newton) will be measured under universal testing machine | Immediately after intervention
  fracture resistance of endodontically treated teeth which were restored with contemporary core buildup materials.

CONTACTS AND LOCATIONS:
Locations (1):
- DIKIOHS, Karachi, Sindh, Pakistan